CLINICAL TRIAL: NCT06802770
Title: Evaluation of Depression and Anxiety Levels of Parents of Children with Spina Bifida
Status: Active, not recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: MAR.UAD.0013
Record Dates: First submitted 2024-12-23; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Spina Bifida
Keywords: spina bifida; anxiety; depression
MeSH Terms: conditions — Spinal Dysraphism; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Spina Bifida Group: Parents ( mother or father) have child with spina bifida
  Interventions: Diagnostic Test: Anxiety, Depression levels

INTERVENTIONS:
Diagnostic Test: Anxiety, Depression levels — Parents of children with spina bifida will be filled out symptom scores regarding depression and anxiety levels.

SUMMARY:
Studies in the literature have measured the anxiety and depression levels of parents of children with spina bifida. Additionally, it has been reported that parents of children with non-neurogenic lower urinary tract dysfunction, such as nocturnal enuresis and overactive bladder, have increased levels of anxiety and depression. In this study, the investigators aim to evaluate, for the first time, the effect of urinary system symptoms and findings in children with spina bifida on the anxiety and depression levels of their parents.

DETAILED DESCRIPTION:
Between January 2024 and December 2024, the demographic data of patients with spina bifida under follow-up, as well as the results of dimercaptosuccinic acid (DMSA) static renal scintigraphy, urinary ultrasonography (USG), and voiding cystourethrography (VCUG), which indicate upper urinary tract (UUT) damage, were recorded. Symptom scoring was performed on the primary caregiver of the child, and anxiety and depression scores were calculated. The Hospital Anxiety and Depression Scale (HADS) and the Beck Anxiety Inventory were used to assess these symptoms in the parents. The presence of renal scarring, hydronephrosis, or vesicoureteral reflux (VUR) in the DMSA was considered as UUT damage. Patients were divided into subgroups based on demographic data, UUT damage, history of febrile urinary tract infections (UTIs), incontinence, and the presence of motor deficits. These groups were then compared in terms of anxiety and depression scores.

ELIGIBILITY:
Inclusion Criteria:

- Having a child with spina bifida

Exclusion Criteria:

- Diagnosis of psychiatric illness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents whom have a child with spina bifida
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety Level- Hospital Anxiety Scale | Baseline
  For Anxiety Hospital Anxiety scale used
  In the Hospital Anxiety Score, the minimum score is 0, and the maximum score is 21. As the score increases, it indicates higher levels of anxiety.
Depression Level | Baseline
  For Depression Hospital Depression scale used
  In the Hospital Depression Score, the minimum score is 0, and the maximum score is 21. As the score increases, it indicates higher levels of depression.
Anxiety Level- BECK Scale | Baseline
  In the BECK Scale, the minimum score is 0, and the maximum score is 63. As the score increases, it indicates higher levels of pain.

CONTACTS AND LOCATIONS:
Overall Officials: CAGRI A. SEKERCİ, Study Director — MARMARA UNİVERSİTY SCHOOL OF MEDİCİNE DEPARTMENT OF UROLOGY
Locations (1):
- Marmara University School of Medicine Urology Department, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided